CLINICAL TRIAL: NCT06176625
Title: Prospective Initiative to Examine and Address Hearing Loss, Vision Loss, and Delirium in a Hospital Setting
Brief Title: Sight and Hearing Investigation Into Effects on Delirium
Acronym: SHIELD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00306862; 1K23AG065443-01 (NIH)
Record Dates: First submitted 2023-12-07; First posted 2023-12-20 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Hearing Loss; Hearing Loss, Age-Related; Hearing Disability; Delirium; Delirium in Old Age; Delirium of Mixed Origin; Delirium With Dementia; Delirium on Emergence; Delirium, Cause Unknown; Delirium Superimposed on Dementia; Delirium Confusional State; Delirium;Non Alcoholic; Hearing Loss, Bilateral; Hearing Loss, Sensorineural; Hearing Loss, Functional; Hearing Loss, High-Frequency; Hearing
MeSH Terms: conditions — Hearing Loss; Presbycusis; Delirium; Emergence Delirium; Confusion; Hearing Loss, Bilateral; Hearing Loss, Sensorineural; Hearing Loss, Functional; Hearing Loss, High-Frequency

STUDY DESIGN:
Intervention Model Description: Initial portion of study is observational in nature.
  For the interventional portion, a baseline period of data collection will first be completed on all three hospital units. Intervention will be initially implemented in one unit and added in each subsequent unit in succession following equivalent time periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Delirium & Sensory Loss (No Intervention): The observational portion of the study, during which participants are screened for delirium. Consented individuals also complete bedside hearing and vision screenings, and provide information regarding care on patient satisfaction questionnaires.
- Baseline Delirium Prevalence (No Intervention): This arm of the interventional portion of the study will be used as baseline comparison data to determine whether implementation of the intervention impacted delirium outcomes. Baseline data collection will be collected for each of the units prior to implementation of the intervention.
- Communication Signage (Active Comparator): For patients who report a little or moderate trouble hearing following the implementation of the intervention, a pink sign will be posted to prompt use of effective communication strategies by nursing staff.
  Interventions: Behavioral: Communication Signage
- Amplifier (Active Comparator): For patients who report a lot of trouble hearing following the implementation of the intervention, a blue sign will be posted to prompt nursing staff to remind patient to make use of amplifier provided as part of the study.
  Interventions: Behavioral: Communication Signage; Behavioral: Amplifier Use

INTERVENTIONS:
Behavioral: Communication Signage — Signage regarding effective communication strategies posted on door to patient's room.
  Arms: Amplifier; Communication Signage
Behavioral: Amplifier Use — Patient is provided amplification device and signage regarding effective communication strategies with reminder to utilize the amplification device posted on door to patient's room.
  Arms: Amplifier

SUMMARY:
The goal of this observational study is to learn about sensory loss in hospital patients with delirium. The main questions it aims to answer are:

* Are hearing and vision loss related to increased risk of having delirium?
* Do hearing and vision loss contribute to more severe delirium?
* Do sensory loss and/or delirium affect patient satisfaction with hospital care?

Participants will be asked to:

* answer delirium screening questions,
* undergo hearing & vision screenings, and
* complete questionnaires about the hospital stay.

The second part of this study is a clinical trial. Researchers will compare different hospital units to see if changing communication affects the number of patients with delirium. The main questions it aims to answer are:

• Does sharing information about communication and/or providing hearing devices change the number of hospital patients with delirium?

Participants in the study will be asked to complete delirium screenings and answer questions about their hearing and communication.

DETAILED DESCRIPTION:
This is a prospective cohort study entitled Sight & Hearing Investigation into Effects on Delirium (SHIELD), which aims of to characterize the impact of sensory impairment (i.e., vision and/or hearing loss) on inpatient delirium and experience. The initial phase of this research includes delirium, hearing, and vision screenings, as well as questionnaires regarding satisfaction with care, all of which are observational and do not constitute treatment or intervention. Researchers will conduct electronic medical record reviews to determine whether new patients have been admitted to the units of recruitment on a daily basis and collect relevant demographic and medical information. Eligible patients will be screened to with the 4AT identify delirium and the 3D-CAM-S to characterize delirium severity. After obtaining informed consent, patients will undergo bedside hearing and vision screenings, and complete patient satisfaction questionnaires.

The second phase of present study aims to determine the impact of improving communication on delirium in the hospital setting. Screenings will be used to identify delirium and measure severity and patients will be asked to report subjective hearing difficulty. Subsequent intervention will involve addressing communication barriers posed by hearing loss by providing training to clinical nursing staff, reinforcing strategies for effective communication through the use of posted signs, and providing amplification devices to eligible patients.

ELIGIBILITY:
Inclusion Criteria:

* inpatient on Johns Hopkins Bayview Medicine A, Medicine B, or Carol Ball unit
* communicates using speech and language
* able to converse in English

Exclusion Criteria:

* nonverbal
* unable to communicate using English language
* currently under airborne or droplet isolation precautions

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1543 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Delirium as Assessed by 4AT Rapid Clinical Test for Delirium (4AT) | Approximately daily during hospitalization up to 6 months
  Diagnosis of delirium using 4AT Rapid Clinical Test for Delirium (4AT). This test has a score range of 0 to 12, with a score of 4 or more indicating a positive delirium result. A score between 1 and 3 is indicative of possible cognitive impairment. Delirium symptom severity can be informally inferred from the test score, but the study will not be using the 4AT Rapid Clinical Test for Delirium (4AT) to measure delirium severity.
Number of Participants with Delirium as Assessed by 4AT Rapid Clinical Test for Delirium in Proportion to Total Number of Patients Screened | Approximately daily during hospitalization up to 6 months
  Counts of delirium diagnosed using 4AT Rapid Clinical Test for Delirium (4AT) score of 4 or greater, in comparison to the total number of patients screened.
  The 4AT Rapid Clinical Test for Delirium (4AT) has a score range of 0 to 12, with a score of 4 or more indicating a positive delirium result. A score between 1 and 3 is indicative of possible cognitive impairment. Delirium symptom severity can be informally inferred from the test score, but the study will not be using the 4AT Rapid Clinical Test for Delirium (4AT) to measure delirium severity.

SECONDARY OUTCOMES:
Severity of Delirium Quantified by the 3-Minute Diagnostic Interview for Confusion Assessment Method-Defined Delirium (3D-CAM) | Approximately daily during hospitalization up to 6 months
  Study participants who score a 1 or higher on the 4AT Rapid Clinical Test for Delirium (4AT) over the duration of time inpatient on the three hospital units of recruitment (Johns Hopkins Bayview Medicine A, Medicine B, and Carol Ball units).
  Quantification of delirium severity from 3-Minute Diagnostic Interview for Confusion Assessment Method-Defined Delirium Severity (3D-CAM-S) score. The possible range of scores is from 0 to 20, with a larger number indicating the presence of more delirium signs and symptoms. However, the diagnosis of delirium using this metric depends on the presence of four characteristic features of delirium.
Satisfaction with Care Assessed Using the Questionnaire on the Quality of Physician-Patient Interaction (QQPI) | Once during hospitalization up to 6 months
  Self-reported satisfaction with hospital care from scores on Questionnaire on the Quality of Physician-Patient Interaction (QQPPI) and/or Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) measures.
  Possible scores on the QQPPI range from 14 to 70; higher scores indicate higher patient satisfaction.
Satisfaction with Care Assessed Using the Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) | Once during hospitalization up to 6 months
  Self-reported satisfaction with hospital care from scores on Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) measures.
  Possible scores on the HCAHPS range from 11 to 62 regarding the hospital stay and between 1 and 5 on each of the two personal health questions. A higher score is consistent with better patient satisfaction and better subjective ratings of personal overall and mental health.

OTHER OUTCOMES:
Hearing Sensitivity as Quantified with Four-Frequency Pure Tone Average (PTA) for the Better-Hearing Ear | Once during hospitalization up to 6 months
  Hearing sensitivity will be quantified based on the average of thresholds measured for four pure tone frequencies (500, 1000, 2000, and 4000 Hz). Thresholds will be measured under earphones during an iPad-based SHOEBOX audiometric screening. PTA values range from -20 to 90 decibels hearing level (dB HL). A higher pure tone average (PTA) suggests that higher signal intensities were necessary for the participant to hear and respond to the stimuli, which also suggests poorer hearing.
  World Health Organization categories for PTA are include 25 or less: no impairment, 26 to 40: slight impairment, 41 to 60: moderate impairment, 61 to 80: severe impairment, and 81 or greater: profound impairment including deafness.
Binocular Distance Visual Acuity Quantified with E-Book from National Health and Aging Trends Study (NHATS) | Once during hospitalization up to 6 months
  Vision screenings will be performed using the National Health and Aging Trends Study (NHATS) Vision e-book developed by Ridgevue Vision on an iPad. Participants will not use glasses or contacts during the testing.
  Distance visual acuity will be measured at 5 feet. Scores range from 50/20 to 4/20, with smaller numbers indicating better distance visual acuity.
Binocular Contrast Sensitivity Quantified with E-Book from National Health and Aging Trends Study (NHATS) | Once during hospitalization up to 6 months
  Vision screenings will be performed using the National Health and Aging Trends Study (NHATS) Vision e-book developed by Ridgevue Vision on an iPad. Participants will not use glasses or contacts during the testing.
  Contrast sensitivity will also be measured at a distance of 5 feet. Scores for this test range from 0.5 to 2.0 with a larger score indicating better contrast sensitivity.
Binocular Near Visual Acuity Quantified with E-Book from National Health and Aging Trends Study (NHATS) | Once during hospitalization up to 6 months
  Vision screenings will be performed using the National Health and Aging Trends Study (NHATS) Vision e-book developed by Ridgevue Vision on an iPad. Participants will not use glasses or contacts during the testing.
  Near visual acuity will be measured at usual reading distance. Scores for this test range from 32/20 to 2.5/20, with smaller numbers indicating better near visual acuity.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas S Reed, Au.D., Ph.D., Principal Investigator — Assistant Professor, Department of Epidemiology; Esther Oh, MD, Ph.D., Principal Investigator — Associate Professor, Departments of Medicine and Psychiatry
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Limited data sets of information may be available to other researchers, pending approval of the Johns Hopkins Medicine Institutional Review Board.
  For participants who have provided informed consent, this information includes demographics (age, sex, race), Charlson comorbidity index score, delirium screening and severity results, hearing screening results, vision screening results, and patient satisfaction data.
  For patients who qualified for study inclusion under waivers of documentation of informed consent and HIPAA, this information includes demographics (age, sex, race) and delirium screening and severity results.

REFERENCES:
- [Background] Pandhi N, Schumacher JR, Barnett S, Smith MA. Hearing loss and older adults' perceptions of access to care. J Community Health. 2011 Oct;36(5):748-55. doi: 10.1007/s10900-011-9369-3. PMID 21301940
- [Background] Reed NS, Boss EF, Lin FR, Oh ES, Willink A. Satisfaction With Quality of Health Care Among Medicare Beneficiaries With Functional Hearing Loss. Med Care. 2021 Jan;59(1):22-28. doi: 10.1097/MLR.0000000000001419. PMID 32925460
- [Background] Mick P, Foley DM, Lin FR. Hearing loss is associated with poorer ratings of patient-physician communication and healthcare quality. J Am Geriatr Soc. 2014 Nov;62(11):2207-9. doi: 10.1111/jgs.13113. No abstract available. PMID 25413192
- [Background] Genther DJ, Betz J, Pratt S, Martin KR, Harris TB, Satterfield S, Bauer DC, Newman AB, Simonsick EM, Lin FR; Health, Aging and Body Composition Study. Association Between Hearing Impairment and Risk of Hospitalization in Older Adults. J Am Geriatr Soc. 2015 Jun;63(6):1146-52. doi: 10.1111/jgs.13456. Epub 2015 Jun 11. PMID 26096388
- [Background] Reed NS, Assi L, Horiuchi W, Hoover-Fong JE, Lin FR, Ferrante LE, Inouye SK, Miller Iii ER, Boss EF, Oh ES, Willink A. Medicare Beneficiaries With Self-Reported Functional Hearing Difficulty Have Unmet Health Care Needs. Health Aff (Millwood). 2021 May;40(5):786-794. doi: 10.1377/hlthaff.2020.02371. PMID 33939509
- [Background] Lin FR, Niparko JK, Ferrucci L. Hearing loss prevalence in the United States. Arch Intern Med. 2011 Nov 14;171(20):1851-2. doi: 10.1001/archinternmed.2011.506. No abstract available. PMID 22083573
- [Background] Congdon N, O'Colmain B, Klaver CC, Klein R, Munoz B, Friedman DS, Kempen J, Taylor HR, Mitchell P; Eye Diseases Prevalence Research Group. Causes and prevalence of visual impairment among adults in the United States. Arch Ophthalmol. 2004 Apr;122(4):477-85. doi: 10.1001/archopht.122.4.477. PMID 15078664
- [Background] Swenor BK, Ramulu PY, Willis JR, Friedman D, Lin FR. The prevalence of concurrent hearing and vision impairment in the United States. JAMA Intern Med. 2013 Feb 25;173(4):312-3. doi: 10.1001/jamainternmed.2013.1880. No abstract available. PMID 23338042
- [Background] Lin FR, Yaffe K, Xia J, Xue QL, Harris TB, Purchase-Helzner E, Satterfield S, Ayonayon HN, Ferrucci L, Simonsick EM; Health ABC Study Group. Hearing loss and cognitive decline in older adults. JAMA Intern Med. 2013 Feb 25;173(4):293-9. doi: 10.1001/jamainternmed.2013.1868. PMID 23337978
- [Background] Hwang PH, Longstreth WT Jr, Thielke SM, Francis CE, Carone M, Kuller LH, Fitzpatrick AL. Longitudinal Changes in Hearing and Visual Impairments and Risk of Dementia in Older Adults in the United States. JAMA Netw Open. 2022 May 2;5(5):e2210734. doi: 10.1001/jamanetworkopen.2022.10734. PMID 35511175
- [Background] Fong TG, Tulebaev SR, Inouye SK. Delirium in elderly adults: diagnosis, prevention and treatment. Nat Rev Neurol. 2009 Apr;5(4):210-20. doi: 10.1038/nrneurol.2009.24. PMID 19347026
- [Background] Witlox J, Eurelings LS, de Jonghe JF, Kalisvaart KJ, Eikelenboom P, van Gool WA. Delirium in elderly patients and the risk of postdischarge mortality, institutionalization, and dementia: a meta-analysis. JAMA. 2010 Jul 28;304(4):443-51. doi: 10.1001/jama.2010.1013. PMID 20664045
- [Background] Harithasan D, Mukari SZS, Ishak WS, Shahar S, Yeong WL. The impact of sensory impairment on cognitive performance, quality of life, depression, and loneliness in older adults. Int J Geriatr Psychiatry. 2020 Apr;35(4):358-364. doi: 10.1002/gps.5237. Epub 2019 Dec 5. PMID 31736109
- [Background] Deal JA, Albert MS, Arnold M, Bangdiwala SI, Chisolm T, Davis S, Eddins A, Glynn NW, Goman AM, Minotti M, Mosley T, Rebok GW, Reed N, Rodgers E, Sanchez V, Sharrett AR, Coresh J, Lin FR. A randomized feasibility pilot trial of hearing treatment for reducing cognitive decline: Results from the Aging and Cognitive Health Evaluation in Elders Pilot Study. Alzheimers Dement (N Y). 2017 Jun 21;3(3):410-415. doi: 10.1016/j.trci.2017.06.003. eCollection 2017 Sep. PMID 29067347
- [Background] Thompson GP, Sladen DP, Borst BJ, Still OL. Accuracy of a Tablet Audiometer for Measuring Behavioral Hearing Thresholds in a Clinical Population. Otolaryngol Head Neck Surg. 2015 Nov;153(5):838-42. doi: 10.1177/0194599815593737. Epub 2015 Jul 16. PMID 26183518
- [Background] Varadaraj V, Assi L, Gajwani P, Wahl M, David J, Swenor BK, Ehrlich JR. Evaluation of Tablet-Based Tests of Visual Acuity and Contrast Sensitivity in Older Adults. Ophthalmic Epidemiol. 2021 Aug;28(4):293-300. doi: 10.1080/09286586.2020.1846758. Epub 2020 Nov 13. PMID 33185485
- [Background] Bellelli G, Morandi A, Davis DH, Mazzola P, Turco R, Gentile S, Ryan T, Cash H, Guerini F, Torpilliesi T, Del Santo F, Trabucchi M, Annoni G, MacLullich AM. Validation of the 4AT, a new instrument for rapid delirium screening: a study in 234 hospitalised older people. Age Ageing. 2014 Jul;43(4):496-502. doi: 10.1093/ageing/afu021. Epub 2014 Mar 2. PMID 24590568
- [Background] Inouye SK, Kosar CM, Tommet D, Schmitt EM, Puelle MR, Saczynski JS, Marcantonio ER, Jones RN. The CAM-S: development and validation of a new scoring system for delirium severity in 2 cohorts. Ann Intern Med. 2014 Apr 15;160(8):526-533. doi: 10.7326/M13-1927. PMID 24733193
- [Background] Livingston G, Huntley J, Sommerlad A, Ames D, Ballard C, Banerjee S, Brayne C, Burns A, Cohen-Mansfield J, Cooper C, Costafreda SG, Dias A, Fox N, Gitlin LN, Howard R, Kales HC, Kivimaki M, Larson EB, Ogunniyi A, Orgeta V, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care: 2020 report of the Lancet Commission. Lancet. 2020 Aug 8;396(10248):413-446. doi: 10.1016/S0140-6736(20)30367-6. Epub 2020 Jul 30. No abstract available. PMID 32738937
- [Background] Lin FR, Ferrucci L, An Y, Goh JO, Doshi J, Metter EJ, Davatzikos C, Kraut MA, Resnick SM. Association of hearing impairment with brain volume changes in older adults. Neuroimage. 2014 Apr 15;90:84-92. doi: 10.1016/j.neuroimage.2013.12.059. Epub 2014 Jan 9. PMID 24412398
- [Background] Cudmore V, Henn P, O'Tuathaigh CMP, Smith S. Age-Related Hearing Loss and Communication Breakdown in the Clinical Setting. JAMA Otolaryngol Head Neck Surg. 2017 Oct 1;143(10):1054-1055. doi: 10.1001/jamaoto.2017.1248. PMID 28837709
- [Background] Pope DS, Gallun FJ, Kampel S. Effect of hospital noise on patients' ability to hear, understand, and recall speech. Res Nurs Health. 2013 Jun;36(3):228-41. doi: 10.1002/nur.21540. Epub 2013 Apr 19. PMID 23606205
- [Background] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Background] Oh ES, Fong TG, Hshieh TT, Inouye SK. Delirium in Older Persons: Advances in Diagnosis and Treatment. JAMA. 2017 Sep 26;318(12):1161-1174. doi: 10.1001/jama.2017.12067. PMID 28973626
- [Background] Marcantonio ER. Delirium in Hospitalized Older Adults. N Engl J Med. 2017 Oct 12;377(15):1456-1466. doi: 10.1056/NEJMcp1605501. PMID 29020579
- [Background] Fick DM, Steis MR, Waller JL, Inouye SK. Delirium superimposed on dementia is associated with prolonged length of stay and poor outcomes in hospitalized older adults. J Hosp Med. 2013 Sep;8(9):500-5. doi: 10.1002/jhm.2077. Epub 2013 Aug 19. PMID 23955965
- [Background] Mohanty S, Gillio A, Lindroth H, Ortiz D, Holler E, Azar J, Boustani M, Zarzaur B. Major Surgery and Long Term Cognitive Outcomes: The Effect of Postoperative Delirium on Dementia in the Year Following Discharge. J Surg Res. 2022 Feb;270:327-334. doi: 10.1016/j.jss.2021.08.043. Epub 2021 Oct 29. PMID 34731730